CLINICAL TRIAL: NCT01282242
Title: MR WITNESS: A Phase IIa Safety Study of Intravenous Thrombolysis With Alteplase in MRI-Selected Patients
Brief Title: A Study of Intravenous Thrombolysis With Alteplase in MRI-Selected Patients
Acronym: MR WITNESS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lee Schwamm (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Lee Schwamm, Vice Chairman, Department of Neurology, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010P001880
Record Dates: First submitted 2011-01-19; First posted 2011-01-24 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-05

CONDITIONS: Acute Stroke
Keywords: acute stroke, IV rt-PA, Activase, Alteplase
MeSH Terms: conditions — Stroke | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IV rt-PA (Experimental): open-label
  Interventions: Drug: IV rt-PA

INTERVENTIONS:
Drug: IV rt-PA — open-label
  Other Names: Alteplase, Activase

SUMMARY:
This study was jointly developed and is jointly led by investigators at Massachusetts General Hospital and the intramural division of NINDS. We are doing this research study to find out if Activase ® (also called alteplase or rt-PA) can safely be given to people with an acute ischemic stroke when their stroke onset was not witnessed making them ineligible for standard thrombolytic (clot busting) therapy. We also want to find out if rt-PA can help people recover better from their stroke.

The purpose of this study is to: 1) see if it is safe to give intravenous (IV) rt-PA to people with unwitnessed stroke but with MRI evidence of early ischemic stroke, 2) see if rt-PA is effective if given to people who are selected for treatment based on MRI evidence of an early stroke, and 3) get information about this new MRI diagnostic methods for guiding stroke treatment.

DETAILED DESCRIPTION:
This study was jointly developed and is jointly led by Massachusetts General Hospital and the NINDS. This is a multi-center, open-label, Phase IIa safety study in adult acute ischemic stroke patients to determine if it is safe to extend intravenous thrombolytic treatment to subjects who are evaluated within 24 hours from last known well ("stroke onset") and eligible to receive thrombolytic treatment within 4.5 hours from symptom discovery with the assistance of an MRI-based "witness" when no human witness of stroke onset is available. The study is designed to investigate the safety in using standard diagnostic MRI in selecting patients for thrombolytic therapy when the last known well time places the patient beyond the current IV thrombolytic time-window.

ELIGIBILITY:
Inclusion Criteria:

* Age, 18 to 85 years inclusive
* Brain MRI findings consistent with early stroke onset
* Clinical diagnosis of acute ischemic stroke with disabling neurological deficit
* Stroke symptoms present for at least 30 minutes with no significant improvement before treatment
* Be last known well (without stroke symptoms) within 24 hours of triage
* Be able to receive IV rt-PA within 4.5 hours from the time the symptoms were discovered.
* MRI diagnostic of acute ischemic stroke and consistent with clinical syndrome
* Time between completion of qualifying MRI studies to treatment initiation ≤ 1 hour

Exclusion Criteria:

* History of intracranial hemorrhage
* Symptoms rapidly improving or only minor before start of study drug.
* Severe stroke as assessed clinically (e.g., NIHSS score >25) or by appropriate imaging techniques (lesion volume > one-third of MCA by visual inspection or >100 cm3 using the ellipsoid estimation formula of ABC/2)
* Stroke or serious head trauma within the previous 3 months
* Administration of heparin within the 48 hours preceding the onset of stroke, with an activated partial-thromboplastin time at presentation exceeding the upper limit of the normal range
* Platelet count of less than 100,000 per cubic millimeter
* Uncontrolled hypertension defined as systolic blood pressure > 185 mm Hg or diastolic blood pressure > 110 mm Hg that cannot be controlled except with continuous parenteral antihypertensive medication
* Blood glucose less than 50 mg per deciliter or greater than 400 mg per deciliter
* Symptoms suggestive of subarachnoid hemorrhage, even if CT/MRI scan was normal
* Oral anticoagulant treatment, regardless of INR.
* Major surgery or severe trauma within the previous 3 months
* Other major disorders associated with an increased risk of bleeding
* Eligible for rt-PA therapy per institutional protocol as part of routine clinical practice
* Non-ischemic etiology demonstrated by neuroimaging
* Neuroimaging (CT or gradient echo MRI) evidence of acute or chronic ICH (non-microbleed)
* Presence of 10 or more microbleeds on GRE (suggestive of amyloid angiopathy)
* Any contraindication for MRI, e.g. presence of a pacemaker, ferromagnetic aneurysm clip, etc, pre-menopausal women with a positive pregnancy blood test, or severe claustrophobia.
* Poor quality MRI- images are not interpretable
* In the opinion of the investigator, the patient is not an appropriate candidate for IV rt-PA
* Women known to be pregnant, lactating or having a positive or indeterminate pregnancy test.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2011-01; Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Schwamm, MD, Principal Investigator — Massachusetts General Hospital; Steven Warach, MD, PhD, Principal Investigator — NINDS/Seton/UT Southwestern Clinical Research Institute of Austin; Ona Wu, PhD, Principal Investigator — Massachusetts General Hospital; Lawrence Latour, PhD, Principal Investigator — NIH Intramural Stroke Program/Suburban Hospital/Washington Hospital Center
Locations (14):
- United States (14):
  - University of Arizona, Tucson, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - NIH/ NINDS, Washington Hospital, Suburban Hospital, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Washington University School of Medicine/Barnes Jewish Hospital, St Louis, Missouri
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Seton/UT Southwestern Medical Center, Austin, Texas
  - Intermountain Healthcare, Murray, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schwamm LH, Wu O, Song SS, Latour LL, Ford AL, Hsia AW, Muzikansky A, Betensky RA, Yoo AJ, Lev MH, Boulouis G, Lauer A, Cougo P, Copen WA, Harris GJ, Warach S; MR WITNESS Investigators. Intravenous thrombolysis in unwitnessed stroke onset: MR WITNESS trial results. Ann Neurol. 2018 May;83(5):980-993. doi: 10.1002/ana.25235. Epub 2018 Apr 27. PMID 29689135
- [Derived] Ali SF, Siddiqui K, Ay H, Silverman S, Singhal A, Viswanathan A, Rost N, Lev M, Schwamm LH. Baseline Predictors of Poor Outcome in Patients Too Good to Treat With Intravenous Thrombolysis. Stroke. 2016 Dec;47(12):2986-2992. doi: 10.1161/STROKEAHA.116.014871. Epub 2016 Nov 10. PMID 27834750

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between January 2011 and February 2016 from 14 sites across the continental United States, and enrolled in 10 of those sites.
Pre-assignment Details: Subjects diagnosed with acute ischemic stroke, last known well within 24 hours of triage and able to receive IV rt-PA within 4.5 hours from symptom discovery based on MRI findings consistent with early stroke onset, were eligible. MRI Signal Intensity Ration values were defined as <1.15 for the primary and <1.25 for the secondary arm of the trial.
Groups:
- Primary SIR <1.15: MRI confirmed early stroke onset, determined by Signal intensity ratio (SIR) <1.15 (SIR = Contralateral Region Of Interest (ROI)/Ipsilateral ROI)
- Secondary SIR <1.25: MRI confirmed early stroke onset, determined by Signal intensity ratio (SIR) <1.25 (SIR = Contralateral Region Of Interest (ROI)/Ipsilateral ROI)
Period: Overall Study
Arm/Group | Primary SIR <1.15 | Secondary SIR <1.25
Started | 80 | 8
Completed | 80 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population consists of all subjects enrolled who suffered an unwitnessed stroke and qualified per AHA guidelines to receive IV tPA within a window of 3-4.5 hours since symptom discovery and whose signal intensity ratio (SIR) on MRI was <1.15 for primary arm and <1.25 for secondary arm.
Groups:
- SIR <1.15: MRI confirmed early stroke onset, determined by Signal intensity ratio (SIR) <1.15 (SIR = Contralateral Region Of Interest (ROI)/Ipsilateral ROI)
- SIR <1.25: MRI confirmed early stroke onset, determined by Signal intensity ratio (SIR) <1.25 (SIR = Contralateral Region Of Interest (ROI)/Ipsilateral ROI)
- Total: Total of all reporting groups
Arm/Group | SIR <1.15 | SIR <1.25 | Total
Number analyzed (Participants) | 80 | 8 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.46 (13.5) | 67.13 (11.63) | 67.43 (13.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 4 | 41
  Male | 43 | 4 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 0 | 6
  Not Hispanic or Latino | 73 | 8 | 81
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 28 | 5 | 33
  White | 47 | 2 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
NIH Stroke Scale (NIHSS) [Mean (Standard Deviation); unit: units on a scale] — NIH Stroke Scale measured the severity of the stroke. The scores ranged between 4 to 42, with higher score indicating worsening of the Outcome. NIHSS score above 20 is indicative of severe stroke.
  units on a scale | 9.31 (5.87) | 10.13 (4.64) | 9.35 (5.91)
Modified Rankin Scale [Mean (Standard Deviation); unit: units on a scale] — Modified Rankin Scale (mRS) measures a subjects degree of disability on a scale of 0 to 6, where 0 is no disability and 6 is death.
  units on a scale | 0.48 (1.09) | 1.38 (2.26) | 1.18 (1.72)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Symptomatic Intracerebral Hemorrhage
Description: Safety of IV rt-PA as evident by rates of symptomatic ICH defined by an increase of 4 points or more on the NIHSS .
Time Frame: Within 7 days from tPA administration.
Measure: Count of Participants; unit: Participants
Groups:
- SIR < 1.25: MRI confirmed early stroke onset, determined by Signal intensity ratio (SIR) <1.25 (SIR = Contralateral Region Of Interest (ROI)/Ipsilateral ROI)
Arm/Group | SIR <1.15 | SIR < 1.25
Number analyzed (Participants) | 80 | 8
Participants | 1 | 1

2. Secondary Outcome: Number of Subjects With Symptomatic Cerebral Edema
Description: Safety of IV rt-PA as evident by rates of symptomatic cerebral edema defined as brain edema with mass effect as the predominant cause of clinical deterioration.
Time Frame: Within 96 hours of tPA administration
Measure: Count of Participants; unit: Participants
Arm/Group | SIR <1.15 | SIR < 1.25
Number analyzed (Participants) | 80 | 8
Participants | 3 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time subjects were consented through study completion, a 90 day period, about 3 months.
Arm/Group | SIR <1.15 | SIR <1.25
All-Cause Mortality (participants affected / at risk) | 7/80 | 1/8
Serious Adverse Events (participants affected / at risk) | 22/80 | 5/8
Other Adverse Events (participants affected / at risk) | 56/80 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SIR <1.15 (N=80) | SIR <1.25 (N=8)
Asthenia (General disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 3 | 0
Brain Oedema (Nervous system disorders) | 6 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0
Cerebral Heamorrhage (Nervous system disorders) | 2 | 1
Cerebrovascular Accident (Nervous system disorders) | 3 | 1
Confusional State (Psychiatric disorders) | 2 | 0
Convulsion (Nervous system disorders) | 2 | 0
Death (General disorders) | 3 | 0
Gastrointestinal Heamorrhage (Gastrointestinal disorders) | 1 | 0
Heamatoma (Vascular disorders) | 1 | 0
Haemorrhage Intracranial (Nervous system disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 1 | 0
Mental Status Changes (Psychiatric disorders) | 2 | 0
Neurological Symptom (Nervous system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Septic Shock (Infections and infestations) | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
ANGIOEDEMA (Vascular disorders) | 0 | 1
BRAIN HERNIATION (Nervous system disorders) | 0 | 1
CAROTID ARTERY STENOSIS (Vascular disorders) | 0 | 1
FALL (Injury, poisoning and procedural complications) | 0 | 1
MYOCARDIAL INFARCTION (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SIR <1.15 (N=80) | SIR <1.25 (N=8)
Agitation (Psychiatric disorders) | 4 | 0
Cerebral Haemorrhage (Nervous system disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 7 | 1
Depression (Psychiatric disorders) | 4 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 5 | 0
Heamorrhagic Transformation (Nervous system disorders) | 18 | 1
Headache (Nervous system disorders) | 13 | 0
Nausea (Gastrointestinal disorders) | 8 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 4 | 2
Pyrexia (General disorders) | 8 | 0
Urinary Tract Infection (Infections and infestations) | 12 | 0
Vomiting (Gastrointestinal disorders) | 6 | 0
Amnesia (Nervous system disorders) | 0 | 1
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ATRIAL FIBRILLATION (Vascular disorders) | 0 | 1
GINGIVAL BLEEDING (General disorders) | 0 | 1
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1
INJECTION SITE EXTRAVASATION (Skin and subcutaneous tissue disorders) | 1 | 1
LIMB INJURY (Injury, poisoning and procedural complications) | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 1
OROPHARYNGEAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This was a single arm open label trial. Genetech provided alteplase free of charge for this NINDS sponsored study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No